CLINICAL TRIAL: NCT03544762
Title: Correlation of 16α-[18F]Fluoro-17β-estradiol PET Imaging With ESR1 Mutation for Prognosis Prediction and Response Evaluation of Hormone Therapy in Primary and Metastatic Breast Cancer
Brief Title: Correlation of 16α-[18F]Fluoro-17β-estradiol PET Imaging With ESR1 Mutation
Acronym: breast
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201512142MINA
Record Dates: First submitted 2018-05-22; First posted 2018-06-04 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer
Keywords: breast cancer; PET; [18F]FES; estrogen receptor; hormone treatment; personalized cancer care
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-FES PET (Experimental): PET/CT
  Interventions: Drug: 18F-FES PET

INTERVENTIONS:
Drug: 18F-FES PET — 18F-FES PET will be performed for each patient. All patients will receive intravenously injection of 5-8 mCi (185-296 MBq) of 18F-FES. PET imaging will be performed on PET/CT system. The 1-frame dynamic data acquisition of thoracic region including the primary tumor will be started immediately after tracer injection. Whole-body PET acquisition from skull base to upper thigh will be started 60 minutes after tracre injection.

SUMMARY:
The propose of this prospective study focuses on the role of [18F]FES PET imaging in patients with breast cancer who might receive or are receiving hormone therapy. First, we will develop and optimize the radiosynthesis and quality control tests of [18F]FES in conditions that meet good manufacturing practice (GMP) requirements. Secondly, patients with or without metastatic breast cancer will be enrolled for the conduction of human study. [18F]FES PET imaging will be performed on patients before the initiation of hormone therapy to predict the prognosis and therapeutic response to hormone therapy. The [18F]FES PET results will be compared with ER status obtained by immunohistochemical (IHC) staining on surgically obtained specimens. Moreover, in patients with progression of metastatic disease, the [18F]FES PET will be correlated with ESR1 gene mutation, which is one of the mechanisms for resistance to hormone therapy.

DETAILED DESCRIPTION:
Breast cancer is the fourth leading cancer death both in female and general population in Taiwan. Breast cancer is a cancer with heterogeneous subtypes, based on gene expression profiles and clinicopathological characteristics. Estrogen receptors (ER) expression of breast cancer has significant prognostic values and determines candidate patients for hormone therapy in both adjuvant and metastatic situations. However, ER expression may be variable within the regions of the tumor or discordant between primary and metastatic lesions. Furthermore, ER expression can change over time along the progression of the disease. Many patients receiving hormone therapy finally develop resistance to hormone therapy despite of ER positive result on prior pathologic specimens. Recently, the mutation of ER-related gene ESR1 has been reported to be associated with the mechanism of development of endocrine resistance.

To assist breast cancer treatment, accurate method for patient selection and response prediction to endocrine and other targeted therapy are required. 16α-[18F]fluoro-17β-estradiol ([18F]FES) is currently the only ER-targeted PET agent validated in previous clinical trials. With the development of [18F]FES PET imaging, the status of ER expression could be detected ER status of tumor cell in vivo without the need of an invasive biopsies.

The propose of this prospective study focuses on the role of [18F]FES PET imaging in patients with breast cancer who might receive or are receiving hormone therapy. First, we will develop and optimize the radiosynthesis and quality control tests of [18F]FES in conditions that meet good manufacturing practice (GMP) requirements. Secondly, patients with or without metastatic breast cancer will be enrolled for the conduction of human study. [18F]FES PET imaging will be performed on patients before the initiation of hormone therapy to predict the prognosis and therapeutic response to hormone therapy. The [18F]FES PET results will be compared with ER status obtained by immunohistochemical (IHC) staining on surgically obtained specimens. Moreover, in patients with progression of metastatic disease, the [18F]FES PET will be correlated with ESR1 gene mutation, which is one of the mechanisms for resistance to hormone therapy.

[18F]FES PET is proposed to be served as an interval assessment tool to evaluate the dynamic changes of ER status in patients receiving hormone therapy. Also, the results of this study will demonstrate the impact of [18F]FES PET as a non-invasive tool on decision making of hormone therapy of breast cancer in addition to IHC stain and ESR1 mutation genetic test. After finishing this project, the non-invasive [18F]FES PET imaging will be proved the potential for the improvement of personalized cancer care.

ELIGIBILITY:
Inclusion Criteria:

* Female patients more than twenty years old
* Patients with breast cancer proven by pathology or cytology
* ER status evaluated by immunohistochemical (IHC) staining; Her2 status evaluated by IHC or in-situ hybridization (ISH)
* Patients will receive hormone therapy as adjuvant therapy or treatment of metastatic disease
* Patients with ESR1 gene analysis
* Life expectancy >3 months.
* ECOG performance status 0 to 2
* Hematologic Function：

  1. Neutrophil count ≥1.5×109/L
  2. Platelet count ≥100×109/L
  3. Hemoglobin ≥9.0 g/dL
* Liver Function：

  1. Total bilirubin level ≤ 1.5 mg/dL
  2. Aspartate transaminase (AST) ≤ 77.5 U/L
  3. alanine transaminase (ALT) ≤ 102.5 U/L
  4. (1) Albumin > 25 g/dL
* Renal Function：Creatinine ≤ 2.0 mg/dL

Exclusion Criteria:

* Patients with known secondary malignancy other than breast cancer
* Patients not suitable for hormone therapy after clinical assessment
* Patients who received neoadjuvant chemotherapy, radiation or hormone therapy before the operation of newly diagnosed breast cancer
* Patients treated with oral or intravenous cytotoxic agent(s) during the same period of hormone therapy
* Pregnant or planning pregnant woman
* Unclear consciousness
* Allergy to drug
* Cannot accept 18F-FES PET
* Breastfeeding
* There are other tumors
* By doctor evaluation to unsuitable

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-09-08 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
PET imaging | in 3 days
  Visual interpretation will be performed first by two independent readers to record if there is any abnormal 18F-FES accumulation. The presence, number, size, character, and location of suspected lesions will be filed for each patient in this study. The final results will be validated by tissue proof, correlation with other imaging, or follow-up results. Semi-quantitative analysis will be performed for each lesion suspected during visual interpretation. Standardized uptake values (SUV) will be obtained by placing regions of interest (ROIs) around the lesions that are identified on visual analysis. The maximum SUV (SUVmax) will be recorded.
  Volumetric parameters will be performed by placing volume of interests (VOIs) around the suspected lesions. VOIs will be generated using defined fix SUV thresholds or algorithm-generated isocontours. Manual adjustment of VOIs is allowed when non-tumoral tissue is incorrectly included by automatic method.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No